CLINICAL TRIAL: NCT03785561
Title: Effect of Research Participation vs. Usual Clinical Treatment on Pain in Patients With Musculoskeletal Disorders: Protocol for a Prospective Cohort Study
Brief Title: Effect of Research Participation Versus Usual Clinical Treatment on Pain in Patients With Musculoskeletal Disorders
Status: Completed | Type: Observational
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Principal Investigator, Marius Henriksen, PT, PhD, Professor, Frederiksberg University Hospital
Other Study IDs: Study participation MSK
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2022-08

CONDITIONS: Musculoskeletal Diseases; Osteoarthritis, Knee; Illness Perceptions
Keywords: Musculoskeletal Diseases; Osteoarthritis, Knee; cohort study; illness perceptions
MeSH Terms: conditions — Musculoskeletal Diseases; Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Exposed (intervention) group: Patients diagnosed with a musculoskeletal disorder, who are currently participating in a health research study at the outpatient osteoarthritis clinic at Frederiksberg Hospital.
  Interventions: Other: participation in a health research study
- Unexposed (comparator) group: The unexposed group is defined as patients, diagnosed with a musculoskeletal disorder receiving standard clinical care at the outpatient osteoarthritis clinic at Bispebjerg and Frederiksberg Hospital. They are not currently enrolled in a health research study concerning their musculoskeletal disorder at Bispebjerg and Frederiksberg Hospital

INTERVENTIONS:
Other: participation in a health research study — Patients diagnosed with a musculoskeletal disorder, who are currently participating in a health research study at the outpatient osteoarthritis clinic at Frederiksberg Hospital
  Groups: Exposed (intervention) group

SUMMARY:
This study explores the effects on pain, function and illness perceptions, of participating in clinical research versus being treated with standard care in patients with musculoskeletal disorders.

DETAILED DESCRIPTION:
Musculoskeletal (MSK) disorders are a major burden on individuals, health systems, and social care systems. Increases in life expectancy and ageing populations are expected to make MSK disorders one of the leading causes of disability by the year 2020.

When faced with a potentially life changing diagnosis of a chronic disease, people (in general) develop an organized pattern of perceptions about their condition, and how it impacts their lives and often, the essentially same stressful event may cause significant variations in perceptions. These different perceptions and coping strategies might affect the way the individual chooses to handle the disease and seek health care assistance, which altogether eventually may affect the course of the illness.

Study participation besides reassurance, could be hypothesized to induce beneficial outcomes for the patients, but is it reasonable to expect an effect of study participation regardless of study intervention, design and group allocation? And is an eventual effect mainly derived from the intervention or from the participants being a selected group?

It remains to be clarified, whether and how study participation affects the individual's treatment effect and perceptions of the illness.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Diagnosed with a musculoskeletal disorder
* Currently enrolled in a health research study hosted by the outpatient osteoarthritis clinic at Frederiksberg Hospital OR Being treated in the outpatient osteoarthritis clinic at Frederiksberg Hospital and not participating in a health research study
* Reads and speaks Danish
* Consents to participation in this survey

Exclusion Criteria:

• We have no formal exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be based on a prospectively sampled cohort of patients from the outpatient osteoarthritis clinic at Frederiksberg Hospital (approximately 1100 patients per year). The OA clinic receives patients with all different kinds of musculoskeletal disorders - not only OA (e.g. rheumatic -, degenerative- and inflammatory disorders in the musculoskeletal system). Patients are identified and will be recruited as they come to the outpatient clinic as part of any health research study or as patients not currently participating in a health research study.
Sampling Method: Non-Probability Sample
Enrollment: 1850 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The Brief Pain Inventory short form | At baseline and end of study (<=1 year)
  The BPI measures the intensity of pain experienced within the last 24 hours and how much pain has interfered with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others, and sleep. In this study we will use the short version (BPI-SF). The BPI-SF is based on numerical rating scales (0-10). The arithmetic mean of the four severity items can be used as measures of pain severity. A lower score indicates less pain interference

SECONDARY OUTCOMES:
PainDETECT questionnaire | At baseline and end of study (<=1 year)
  PainDETECT questionnaire was developed to detect neuropathic pain components in adult patients. The questionnaire consists of seven questions addressing the quality of neuropathic pain symptoms; it is completed entirely by the patient. It contains seven questions that address the quality of neuropathic pain symptoms scored from 0 to 5 (never = 0, hardly noticed = 1, slightly = 2; moderately = 3, strongly = 4, very strongly = 5), four questions addressing the pain course pattern (scored from -1 to +1) and one question concerning radiation of pain into other parts of the body (yes (+2)/no (0)). The final score between -1 and 38 indicates the likelihood of a neuropathic pain component. A score of ≤ 12 indicates that pain is unlikely to have a neuropathic component, while a score of ≥ 19 suggests that pain is likely to have a neuropathic component
The Brief Illness Perception Questionnaire | At baseline and end of study (<=1 year)
  The Brief illness perception questionnaire BIPQ is a generic questionnaire developed to measure illness perception in a variety of illnesses. The questionnaire is patient-reported and assesses perceptions on the following five dimensions: Identity, Cause, Timeline, Consequences and Cure-Control. It contains eight numerical rating scales questions (0-10) and a memo field based on the patients' own beliefs about their condition. In some circumstances it may be possible to compute an overall score which represents the degree to which the illness is perceived as threatening or benign. To compute the score, reverse score items 3, 4, and 7 and add these to items 1, 2, 5, 6, and 8. A higher score reflects a more threatening view of the illness.
Widespread Pain Index | At baseline and end of study (<=1 year)
  Guided by a drawing the participants indicate each area that they have felt pain in over the last week. Pain due to other known illnesses should be excluded from the assessment. There are 19 areas and the index ranges from 0 - 19, with 19 being worst. The WPI is used as part of the ACR fibromyalgia classification criteria but can be used for other pain related disorders
EQ-5D-3L | At baseline and end of study (<=1 year)
  EQ-5D is a standardised measure of health status that provides a simple, generic measure of health. It is applicable to a wide range of health conditions. EQ-5D is designed for self-completion by respondents and is ideally suited for use in postal surveys, in clinics, and in face-to-face interviews and takes only a few minutes to complete. The EQ-5D-3L essentially consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. The EQ VAS records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. This information can be used as a quantitative measure of health outcome as judged by the individual respondents
Health Assessment Questionnaire (Disability) | At baseline and end of study (<=1 year)
  HAQ-DI (HAQ-disability) contains 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities. There are 2 or 3 questions for each section. Scoring within each section is from 0 (without any difficulty) to 3 (unable to do). For each section the score given to that section is the worst score within the section, i.e. if one question is scored 1 and another 2, then the score for the section is 2. In addition, if an aide or device is used or if help is required from another individual, then the minimum score for that section is 2. If the section score is already 2 or more then no modification is made. The 8 scores of the 8 sections are summed and divided by 8. If one section is not completed by a subject, then the summed score would be divided by 7. Scores of 0 to 1 are generally considered to represent mild to moderate difficulty, 1 to 2 moderate to severe disability, and 2 to 3 severe to very severe disability

CONTACTS AND LOCATIONS:
Overall Officials: Henning Bliddal, DMSc, Principal Investigator — The Parker institute
Locations (1):
- The Parker Institute, Frederiksberg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
The Capital region of Denmark will normally only accept sharing of anonymous data

REFERENCES:
- [Derived] Ginnerup-Nielsen E, Christensen R, Bliddal H, Henriksen M. Effect of research participation versus usual clinical care in patients with rheumatic and musculoskeletal disorders: a prospective cohort study. RMD Open. 2023 Oct;9(4):e003414. doi: 10.1136/rmdopen-2023-003414. PMID 37797965